CLINICAL TRIAL: NCT00580632
Title: Workload, Clinical and Therapeutic Management of Psoriatic Arthritis
Brief Title: Study Evaluating Workload, Clinical and Therapeutic Management of Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trials Registry Specialist), Wyeth
Other Study IDs: 0881A-102389
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2007-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Spain, there is little data available concerning the evolution and treatment of Psoriatic Arthritis by rheumatologists and dermatologists. This study is designed to obtain more data about the clinical and therapeutic management of Psoriatic Arthritis in Dermatology and Rheumatology Medical centers.

ELIGIBILITY:
Inclusion Criteria:

1. patients older than 18 years with a psoriatic arthritis diagnosis that go to dermatologic and/or rheumatologic centers or primary care centers.
2. patients that receive pharmacologic treatment for their condition
3. patients that give their written consent to participate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriatic Arthritis Patients with a representative geographic sample
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine diagnosis and evolution time of patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer